CLINICAL TRIAL: NCT01268332
Title: Expanded Safety and Adherence Study of a Non-medicated Intravaginal Ring
Brief Title: Safety and Adherence of a Non-medicated Intravaginal Ring (IVR)
Acronym: MTN-005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); Microbicide Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Population Council #508; NCT00672425 (obsolete NCT alias)
Record Dates: First submitted 2010-12-28; First posted 2010-12-30 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Placebo IVR as a delivery method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravaginal Ring (Experimental): Insertion of intravaginal ring at enrollment. The intravaginal ring should stay in place for 12 consecutive weeks and will be removed by a physician at the Week 12 study visit.
  Interventions: Drug: Non-medicated Intravaginal Ring
- No Intravaginal Ring (No Intervention): Intravaginal ring will not be inserted into participants.

INTERVENTIONS:
Drug: Non-medicated Intravaginal Ring — Cured silicone elastomer composed of an elastomer base, normal propylorthosilicate, and titanium dioxide. The ring will not contain an active pharmaceutical ingredient.
  Other Names: Placebo Intravaginal Ring
  Arms: Intravaginal Ring

SUMMARY:
The purpose of this study is to evaluate the safety of and adherence to a non-medicated IVR in HIV uninfected women over 12 weeks of use.

DETAILED DESCRIPTION:
Women comprise a growing proportion of new HIV infections worldwide. Intravaginal rings (IVRs) used to deliver microbicides have the potential to significantly reduce the heterosexual transmission of HIV if found to be safe, acceptable, and effective against HIV infection. This study will investigate the safety and acceptability of a non-medicated silicone elastomer IVR in sexually active HIV uninfected women.

The expected duration of this study for each participant is 16 weeks. Study participants will be randomly assigned to one of two arms. Participants in Group A will insert an IVR into their vagina at study entry. The IVR will remain in place for 12 weeks until removed by a physician. Follow up will continue for an additional 4 weeks after IVR removal. Participants in Group B will not receive an IVR, but will follow the same study schedule as those in Group A.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* General good health
* Sexually active
* Agree to use an effective method of contraception
* Normal Pap smear result within 12 months prior to study entry
* Agree to not participate in other drug or device research studies for the duration of study participation
* Agree to not use any intravaginal product for the duration of study participation

Exclusion Criteria:

* History of adverse reaction to silicone, latex, or titanium dioxide
* Current male sex partner with known history of adverse reaction to silicone, latex, or titanium dioxide
* Last pregnancy outcome within 30 days or less prior to enrollment
* History of hysterectomy
* Any abnormal pelvic exam finding
* Pregnant
* Condition that, in the opinion of the investigator, would interfere with the study
* Severe pelvic relaxation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2013-03-07 (Actual)

PRIMARY OUTCOMES:
Adherence to intravaginal ring | Throughout study
Grade 2 or higher adverse event | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hoesley, MD, Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Bronx-Lebanon Hospital Center, The Bronx, New York
- National AIDS Research Institute, Pune, India